CLINICAL TRIAL: NCT03778216
Title: Treating Avoidant/Restrictive Food Intake Disorder (ARFID) Using Family-Based Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, James Dale Lock, Principal Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 40043; SPO 125881 (Other Grant/Funding Number: National Eating Disorders Association)
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Avoidant / Restrictive Food Intake Disorder
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FBT-ARFID (Experimental): Family Based Treatment of child ARFID
  Interventions: Behavioral: Family Based Treatment
- Usual Care (No Intervention): Continued usual care for ARFID with the exception of any Family Based Treatment

INTERVENTIONS:
Behavioral: Family Based Treatment
  Other Names: FBT-ARFID
  Arms: FBT-ARFID

SUMMARY:
Although Avoidant/Restrictive Food Intake Disorder (ARFID) was formally introduced in DSM-5, no specialized intervention has yet been empirically studied. This randomized controlled crossover trial (RCCT) will test the feasibility and acceptability of a novel intervention, Family-Based Treatment of Avoidant/Restrictive Food Intake Disorder (FBT-ARFID) for patients ages 5-12 years old.

DETAILED DESCRIPTION:
Potential subjects aged 5 years to 12 years, 11 months old with anorexia nervosa (AN) diagnosed with ARFID and their families will be recruited will be recruited through Stanford University, pediatricians, mental health experts, clinics treating EDs, and local parents' groups. Those eligible for the program will be invited to read and sign informed consent forms and complete the baseline assessment. They will then be randomized to the FBT-ARFID program either immediately after their screening or 3 months after assessment (i.e., to a usual care group). FBT-ARFID consists of 22 sessions over a 6-month period.

There will be 3 major assessment time points for those in the FBT-ARFID Arm: Baseline, 3 months into treatment, and EOT. There will be 4 major assessment time points for those in Usual Care: Baseline, transition to treatment (3 months after the usual care period is complete), 3 months into treatment, and EOT. Both the child and the parent will complete measures at these time points. In addition, patients and parents will participate in ongoing qualitative assessments before treatment (BL), throughout treatment (every other session), and at EOT.

ELIGIBILITY:
Inclusion Criteria:

* children meeting DSM-V criteria for ARFID
* children between the ages of 5 to 12 years old

Exclusion Criteria:

* any medical complications or severe mental disorder (psychosis, low-functioning Autism) that may reduce compliance with the study procedures or require more intensive care to manage the symptoms
* a severe parental mental disorder (e.g., psychotic depression, psychosis, substance dependence)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Estimated Body Weight (EBW) | following 6 months of treatment or 3 months of usual care
  individual with ARFID's body weight at end of condition

SECONDARY OUTCOMES:
Symptom Severity | following 6 months of treatment or 3 months of usual care
  individual with ARFID's symptom severity at end of condition according to the Pica, ARFID, and Rumination Disorder Interview (PARDI). The symptom severity subscale will be used where the higher the score, the greater the ARFID severity. A total of 17 items rated on a scale of 0 to 6 are included in this subscale and the average is reported.

CONTACTS AND LOCATIONS:
Overall Officials: James D Lock, MD, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No